CLINICAL TRIAL: NCT00321672
Title: A Multicenter Randomized, Double-Blind, Controlled Study of NGX-4010 for the Treatment of Painful HIV-Associated Neuropathy
Brief Title: Study of NGX-4010 for the Treatment of Painful HIV-Associated Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NeurogesX (Industry)
Responsible Party: Trudy Vanhove, VP Clinical Development, NeurogesX
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C119
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Results first posted 2011-06-14 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-05

CONDITIONS: Pain; HIV Infections; Peripheral Nervous System Diseases
Keywords: Analgesics; Capsaicin; Neuropathic pain; Neuropathy; Distal sensory polyneuropathy; Peripheral neuropathy; Dermal assessment; Pain measurement
MeSH Terms: conditions — Pain; HIV Infections; Peripheral Nervous System Diseases; Neuralgia | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- NGX-4010, 60 minutes (Experimental)
  Interventions: Drug: NGX-4010, 8% capsaicin patch
- NGX-4010, 30 minutes (Experimental)
  Interventions: Drug: NGX-4010, 8% capsaicin patch
- 0.04% conc. capsaicin patch, 60 min. (Other)
  Interventions: Drug: 0.04% capsaicin patch
- 0.04% conc. capsaicin patch, 30 min. (Other)
  Interventions: Drug: 0.04% capsaicin patch

INTERVENTIONS:
Drug: NGX-4010, 8% capsaicin patch — Up to 4 NGX-4010 patches of 280 cm^2 each were applied to the feet (2 per foot) for 60 minutes.
  Other Names: the brandname of NGX-4010, 8% capsaicin patch is Qutenza.
  Arms: NGX-4010, 60 minutes
Drug: 0.04% capsaicin patch — Up to 4 control patches of 280 cm^2 each were applied to the feet (2 per foot) for 60 minutes.
  Other Names: NGX-4010
  Arms: 0.04% conc. capsaicin patch, 60 min.
Drug: NGX-4010, 8% capsaicin patch — Up to 4 NGX-4010 patches of 280 cm^2 each were applied to the feet (2 per foot) for 30 minutes.
  Other Names: The brandname of NGX-4010, 8% capsaicin patch is Qutenza.
  Arms: NGX-4010, 30 minutes
Drug: 0.04% capsaicin patch — Up to 4 control patches of 280 cm^2 each were applied to the feet (2 per foot) for 30 minutes.
  Other Names: NGX-4010
  Arms: 0.04% conc. capsaicin patch, 30 min.

SUMMARY:
The purpose of the study was to assess the efficacy and safety of NGX-4010 applied for 30 or 60 minutes for the treatment of painful HIV-associated neuropathy.

DETAILED DESCRIPTION:
Study C119 was a multicenter, randomized, double-blind, controlled evaluation of the efficacy and safety of NGX-4010 for the treatment of painful HIV-associated neuropathy. Eligible subjects had painful HIV-associated neuropathy resulting from HIV disease and/or antiretroviral drug exposure in both feet, with average numeric pain rating scale (NPRS) scores during screening of 3 to 9 (inclusive). Up to four patches covering an area of up to 1120 square centimeters could be used during a single treatment administration in this study. Subjects were randomly assigned to receive active NGX-4010 patches (8% capsaicin) or low-concentration control patches (0.04% capsaicin) identical in appearance, at doses (patch application duration) of either 30 or 60 minutes, according to a 2:1:2:1 allocation scheme.

Subjects could be on stable chronic oral pain medication regimens, but could not be using any topical pain medications on the affected areas. NPRS scores for the average pain in the past 24 hours were recorded daily in the evening, beginning on the day of the Screening Visit (usually on Day -14). Subjects continued to record NPRS scores in a take-home diary from the evening on the day of treatment through the evening before the Termination Visit at Week 12. Subjects returned for interim follow-up visits at Weeks 4 and 8 following study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Documented evidence of HIV-1 infection
* Documented diagnosis of painful HIV-associated distal symmetric polyneuropathy resulting from HIV disease and/or antiretroviral drug exposure To be confirmed based on symptoms of pain, burning or dysesthetic discomfort in both feet for at least 2 months prior to Screening Visit, AND absent or diminished ankle reflexes OR at least one of following: distal diminution of vibration sensation or pain or temperature sensation in legs
* Average NPRS scores during screening period of 3 to 9, inclusive
* Life expectancy of 12 months or longer per Investigator's judgment
* Intact, unbroken skin over painful areas to be treated
* If taking chronic pain medications, be on stable regimen for at least 21 days prior to Day 0 and willing to maintain medications at same stable dose(s) and schedule throughout study
* Female subjects with child-bearing potential: negative serum pregnancy test performed at Screening Visit
* Willing to use effective methods of birth control and/or refrain from conception process during study and for 30 days following study drug exposure
* Willing and able to comply with protocol for duration of study

Exclusion Criteria:

* Concomitant opioid medication, unless orally or transdermally administered and not exceeding total daily dose of morphine 80 mg/day or equivalent; parenteral opioids not allowed
* Unavailability of effective rescue medication strategy for subject, such as unwillingness to use opioid analgesics during study treatment or high tolerance to opioids precluding ability to relieve treatment-associated discomfort as judged by investigator
* Active substance abuse or history of chronic substance abuse within past year or prior chronic substance abuse (including alcoholism) judged likely to recur during study period by investigator
* Recent use (within 21 days preceding Day 0) of any topically applied pain medication, such as non-steroidal anti-inflammatory drugs, menthol, methyl salicylate, local anesthetics including Lidoderm® (lidocaine patch 5%), steroids or capsaicin products on painful areas
* Started or stopped treatment with one or more neurotoxic antiretroviral agents (ie, didanosine [ddI], zalcitabine [ddC], or stavudine [d4T] during 8 weeks prior to Day 0
* Participation in previous clinical trial in which subject received either blinded or open-label NGX-4010
* Current use of any investigational agent or Class 1 anti-arrhythmic drugs (such as tocainide and mexiletine)
* Evidence of another contributing cause for peripheral neuropathy, e.g., current uncontrolled diabetes mellitus (HbA1c≥9%) or history of diabetes mellitus preceding onset of HIV-associated neuropathy (HIV-AN); hereditary neuropathy; vitamin B12 deficiency (B12 level ≤200pg/mL at screening); or treatment within 90 days prior to Screening Visit with any drug that may have contributed to sensory neuropathy
* Hypertension, unless adequately controlled by medication
* Significant ongoing pain from other cause(s) that may interfere with judging HIV-AN related pain
* Any implanted medical device for treatment of neuropathic pain
* Hypersensitivity to capsaicin (i.e., chili peppers or over-the-counter (OTC) capsaicin products), local anesthetics, opioid-based oral analgesics or adhesives
* Significant medical conditions (including active malignancy defined as treatment required in last 5 years) that in opinion of investigator would interfere with ability to complete study or evaluation of AEs
* Recent significant medical-surgical intervention that in judgment of Investigator would interfere with ability to complete study or evaluation of AEs; examples include to major surgery, or receipt of immunosuppressive therapy within 3 months prior to Day 0
* Evidence of cognitive impairment including dementia that may interfere with subject's ability to complete daily pain diaries requiring recall of average HIV-associated neuropathy pain level in past 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trudy F Vanhove, MD, Study Director — NeurogesX

REFERENCES:
- [Derived] Brown S, Simpson DM, Moyle G, Brew BJ, Schifitto G, Larbalestier N, Orkin C, Fisher M, Vanhove GF, Tobias JK. NGX-4010, a capsaicin 8% patch, for the treatment of painful HIV-associated distal sensory polyneuropathy: integrated analysis of two phase III, randomized, controlled trials. AIDS Res Ther. 2013 Jan 28;10(1):5. doi: 10.1186/1742-6405-10-5. PMID 23351618
- [Derived] Clifford DB, Simpson DM, Brown S, Moyle G, Brew BJ, Conway B, Tobias JK, Vanhove GF; NGX-4010 C119 Study Group. A randomized, double-blind, controlled study of NGX-4010, a capsaicin 8% dermal patch, for the treatment of painful HIV-associated distal sensory polyneuropathy. J Acquir Immune Defic Syndr. 2012 Feb 1;59(2):126-33. doi: 10.1097/QAI.0b013e31823e31f7. PMID 22067661

RESULTS

PARTICIPANT FLOW:
Groups:
- NGX-4010, 60 Minutes: Treatment with capsaicin patches consisted of a one time application administered at any time of the day on Study Day 0. Subjects were randomized to receive NGX 4010 (high concentration capsaicin, 640 mcg/cm^2) for 60 minutes.
- Control Group, 60 Minutes: Treatment consisted of a one time application administered at any time of the day on Study Day 0. Subjects were randomized to receive a Control patch (low concentration capsaicin, 3.2 mcg/cm^2) for 60 minutes. The low dose of 3.2 mcg/cm^2 (0.04% w/w) used as the Control in this study was selected because it was expected to cause perceptible local sensation, thereby preserving the blind.
- NGX-4010, 30 Minutes: Treatment with capsaicin patches consisted of a one time application administered at any time of the day on Study Day 0. Subjects were randomized to receive NGX 4010 (high concentration capsaicin, 640 mcg/cm^2) for 30 minutes.
- Control Group , 30 Minutes: Treatment consisted of a one time application administered at any time of the day on Study Day 0. Subjects were randomized to receive a Control patch (low concentration capsaicin, 3.2 mcg/cm^2) for 30 minutes. The low dose of 3.2 mcg/cm^2 (0.04% w/w) used as the Control in this study was selected because it was expected to cause perceptible local sensation, thereby preserving the blind.
Period: Overall Study
Arm/Group | NGX-4010, 60 Minutes | Control Group, 60 Minutes | NGX-4010, 30 Minutes | Control Group , 30 Minutes
Started | 165 | 89 (One randomized to 30 minutes received 60 minutes. Under 30 for efficacy and under 60 for safety.) | 167 | 73 (One randomized to 30 minutes received 60 minutes. Under 30 for efficacy and under 60 for safety.)
Completed | 153 | 81 | 156 | 71
Not Completed | 12 | 8 | 11 | 2
Not completed — Withdrawal by Subject | 5 | 1 | 2 | 0
Not completed — Noncompliance | 1 | 2 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 4 | 2
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Too far to travel for visits | 1 | 0 | 0 | 0
Not completed — Incarcerated | 0 | 0 | 2 | 0
Not completed — Moved out of state | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Diagnosis of testicular cancer | 0 | 1 | 0 | 0
Not completed — Extensive travel required for new job | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NGX-4010, 60 Minutes | Control Group, 60 Minutes | NGX-4010, 30 Minutes | Control Group , 30 Minutes | Total
Number analyzed (Participants) | 165 | 90 | 167 | 72 | 494
Age Continuous [Mean (Standard Deviation); unit: years] — 60 minutes control group - one randomized 30 minutes received 60 minutes. Under 30 for efficacy and under 60
  30 minutes control goup, one randomized to 30 minutes received 60 minutes. Under 30 for efficacy and under 60 for safety.
  years | 49.0 (8.52) | 50.1 (9.33) | 50.5 (8.34) | 49.3 (7.78) | 49.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants] — 60 minutes control group - one randomized 30 minutes received 60 minutes. Under 30 for efficacy and under 60
  30 minutes control goup, one randomized to 30 minutes received 60 minutes. Under 30 for efficacy and under 60 for safety.
  Participants
    Female | 17 | 11 | 25 | 9 | 62
    Male | 148 | 79 | 142 | 63 | 432

OUTCOME MEASURES:

1. Primary Outcome: The Primary Measure of Efficacy Was the Percent Change in the "Average Pain for the Past 24 Hours" Numeric Pain Rating Scale (NPRS) Score From Baseline During Weeks 2 to 12.
Description: Efficacy was assessed by daily Numeric Pain Rating Scale (NPRS) capturing "average pain for the past 24 hours" for painful HIV-associated neuropathy area(s) at approximately 9 PM every evening throughout the 12-week study period. The NPRS is an 11-point scale (0 to 10) with 0 indicating no pain and 10 indicating the worst possible pain.
Time Frame: Weeks 2-12
Population: Analyses were intention to treat (ITT). A modified last observation carried forward (LOCF) approach was used to impute missing data. Each NGX-4010 group was compared with its respective control group.
Measure: Least Squares Mean (Standard Error); unit: Percent Change from baseline
Groups:
- NGX-4010 Total: Treatment with capsaicin patches consisted of a one time application administered at any time of the day on Study Day 0. Subjects were randomized to receive NGX 4010 (high concentration capsaicin, 640 mcg/cm^2) for 30 or 60 minutes.
- Control, Total: Treatment consisted of a one time application administered at any time of the day on Study Day 0. Subjects were randomized to receive a Control patch (low concentration capsaicin, 3.2 mcg/cm^2) for 30 or 60 minutes. The low dose of 3.2 mcg/cm^2 (0.04% w/w) used as the Control in this study was selected because it was expected to cause perceptible local sensation, thereby preserving the blind.
Arm/Group | NGX-4010, 60 Minutes | Control Group, 60 Minutes | NGX-4010, 30 Minutes | Control Group , 30 Minutes | NGX-4010 Total | Control, Total
Number analyzed (Participants) | 165 | 90 | 167 | 72 | 332 | 162
Percent Change from baseline | -32.8 (2.41) | -30.0 (3.27) | -26.2 (2.39) | -19.1 (3.61) | -29.5 (1.70) | -24.5 (2.43)
Statistical Analysis 1: Comparison: NGX-4010 Total vs Control, Total; The null hypothesis was that there was no difference between the average percent change in NPRS scores from baseline to weeks 2-12 between the total control and total NGX-4010 groups. The ratio of means between the 30- and 60-minute control group [1.57 (90% CI: 1.12-2.35)] was > than the pre-specified equivalence margin ratio of 80-125%. Hence, the control groups could not be pooled and comparisons were performed between the 30- and 60-minute NGX-4010 groups and their respective control groups; Test type: Superiority or Other; p = 0.0967, ANCOVA — All stastical tests of hypotheses were two-sided and at the 5% level of significance; Treatment differences were compared by a gender stratified analysis of covariance (ANCOVA) model with Baseline pain score as the only covariate
Statistical Analysis 2: Comparison: NGX-4010, 60 Minutes vs Control Group, 60 Minutes; Test type: Superiority or Other; p = 0.4884, ANCOVA — All stastical tests of hypotheses were two-sided and at the 5% level of significance. No multiplicity adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NGX-4010, 30 Minutes vs Control Group , 30 Minutes; Test type: Superiority or Other; p = 0.1031, ANCOVA — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Absolute Change in the Mean "Average Pain for the Past 24 Hours" Numeric Pain Rating Scale (NPRS) Score From Baseline During Weeks 2 to 12.
Time Frame: Weeks 2-12.
Measure: Least Squares Mean (Standard Error); unit: Numeric Pain Rating Scale (0 to 10)
Arm/Group | NGX-4010, 60 Minutes | Control Group, 60 Minutes | NGX-4010, 30 Minutes | Control Group , 30 Minutes | NGX-4010 Total | Control, Total
Number analyzed (Participants) | 165 | 90 | 167 | 72 | 332 | 162
Numeric Pain Rating Scale (0 to 10) | -2.0 (0.15) | -1.8 (0.20) | -1.6 (0.14) | -1.1 (0.22) | -1.8 (0.10) | -1.4 (0.15)
Statistical Analysis 1: Comparison: NGX-4010 Total vs Control, Total; The null hypothesis was: "There is no difference between the total Control and total NGX-4010 in the absolute change in NPRS scores from Baseline during Weeks 2-12."; Test type: Superiority or Other; p = 0.0831, ANCOVA — All statistical tests of hypotheses were two-sided and at the 5% level of significance; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: NGX-4010, 60 Minutes vs Control Group, 60 Minutes; Test type: Superiority or Other; p = 0.4680, ANCOVA — All statistical tests of hypotheses were two-sided and at the 5% level of significance. No multiplicity adjustments were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NGX-4010, 30 Minutes vs Control Group , 30 Minutes; Test type: Superiority or Other; p = 0.0896, ANCOVA — [p-value comment as in outcome 2, analysis 2]; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Proportion of Subjects Reaching 30% Decrease in Their Mean "Average Pain for the Past 24 Hours" Numeric Pain Rating Scale (NPRS) Score From Baseline During Weeks 2 to 12
Time Frame: Weeks 2-12
Measure: Number; unit: Percentage of Participants
Arm/Group | NGX-4010, 60 Minutes | Control Group, 60 Minutes | NGX-4010, 30 Minutes | Control Group , 30 Minutes | NGX-4010 Total | Control, Total
Number analyzed (Participants) | 165 | 90 | 167 | 72 | 332 | 162
Percentage of Participants | 48 | 45 | 39 | 26 | 43 | 36
Statistical Analysis 1: Comparison: NGX-4010 Total vs Control, Total; The null hypothesis was: "There is no difference between the total Control and total NGX-4010 group in the Proportion of Subjects Reaching 30% Decrease in Their Mean "Average Pain for the Past 24 Hours" NPRS Score From Baseline During Weeks 2 to 12."; Test type: Superiority or Other; p = 0.0662, Regression, Logistic — All statistical tests of hypotheses were two-sided and at the 5% level of significance; A logistic regression analysis, with the Baseline NPRS score and gender as covariates, was performed
Statistical Analysis 2: Comparison: NGX-4010, 60 Minutes vs Control Group, 60 Minutes; Test type: Superiority or Other; p = 0.5582, Regression, Logistic — [p-value comment as in outcome 2, analysis 2]; A logistic regression analysis, with the Baseline NPRS score and gender as covariates, was performed
Statistical Analysis 3: Comparison: NGX-4010, 30 Minutes vs Control Group , 30 Minutes; Test type: Superiority or Other; p = 0.0553, Regression, Logistic — [p-value comment as in outcome 2, analysis 2]; A logistic regression analysis, with the Baseline NPRS score and gender as covariates, was performed

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | NGX-4010, 60 Minutes | Control Group, 60 Minutes | NGX-4010, 30 Minutes | Control Group , 30 Minutes | NGX-4010 Total | Control, Total
Serious Adverse Events (participants affected / at risk) | 13/165 | 7/90 | 6/167 | 2/72 | 19/332 | 9/162
Other Adverse Events (participants affected / at risk) | 160/165 | 73/90 | 149/167 | 61/72 | 309/332 | 134/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NGX-4010, 60 Minutes (N=165) | Control Group, 60 Minutes (N=90) | NGX-4010, 30 Minutes (N=167) | Control Group , 30 Minutes (N=72) | NGX-4010 Total (N=332) | Control, Total (N=162)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Giardiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis tuberculous (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Polytraumatism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NGX-4010, 60 Minutes (N=165) | Control Group, 60 Minutes (N=90) | NGX-4010, 30 Minutes (N=167) | Control Group , 30 Minutes (N=72) | NGX-4010 Total (N=332) | Control, Total (N=162)
Application site erythema (General disorders) | 97 (97) | 34 (34) | 79 (79) | 24 (24) | 176 (176) | 58 (58)
Application site pain (General disorders) | 139 (139) | 29 (29) | 135 (135) | 33 (33) | 274 (274) | 62 (62)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (4) | 10 (10) | 2 (2) | 20 (20) | 6 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5) | 7 (7) | 7 (7) | 12 (12) | 12 (12) | 19 (19)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 3 (3) | 4 (4) | 5 (5) | 9 (9)

LIMITATIONS AND CAVEATS:
Differences between the 60- and 30-minute Control groups prevented pooling according to prespecified criteria resulting in treatment comparisons between 60- and 30-minute NGX-4010 groups and their respective Control groups with relatively low power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The PI shall comply with the sponsor's requests to delete references to trade secrets, intellectual properties or other proprietary information.